CLINICAL TRIAL: NCT07234318
Title: Non-interventional Study to Evaluate the Anti-inflammatory Effects and the Clinical Efficacy of Topical Water Free Cyclosporin 0.1% Eye Drops in Patients With Dry Eye Disease and Associated Ocular Surface Inflammation Non-responding to Artificial Tears: the FOCUS Study
Brief Title: Non-interventional Study to Evaluate the Anti-inflammatory Effects and the Clinical Efficacy of Topical Water Free Cyclosporin 0.1% Eye Drops in Patients With Dry Eye Disease and Associated Ocular Surface Inflammation Non-responding to Artificial Tears
Status: Not yet recruiting | Type: Observational
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Other Study IDs: LT10460-401
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Cyclosporin — This medicinal product contains cyclosporine 0.1% as an active ingredient and pefluorobutylpentane as vehicle.

SUMMARY:
The FOCUS study aims to evaluate the clinical efficacy of 0.1% cyclosporine eye drops solution (Vevizye®, Laboratoires THEA) in patients with moderate to severe dry eye disease characterized by ocular surface inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* No patients with other ophthalmic diseases than DED
* Chronic dry eye defined as longer than six months since diagnosis
* OSDI score > 22
* Conjunctival Hyperemia ≥ Grade 3 (Efron Scale)
* Current use of tear substitutes for at least 3 months not to be considered as sufficient by the investigator/treating physician
* Need to add cyclosporine eye drops to tear substitutes as judged by the investigator/treating physician

Exclusion Criteria:

Ophthalmic exclusion criteria

* Far best corrected visual acuity < 1/10
* Severe Dry Eye associated with:

  * Eyelid malposition
  * Stevens Johnson Syndrome
  * Corneal dystrophy
  * Ocular neoplasia
  * Filamentous keratitis
  * Corneal neovascularisation
  * Orbital radiotherapy
  * Dry eye related to Graft Versus Host Disease (GVHD)
* History of any of the following within last 3 months:
* Systemic treatment of dry eye
* Systemic treatment of Meibomian Gland Dysfunction (MGD)
* Isotretinoïde,
* Cyclosporine,
* Tacrolimus, Siromilus, Pimecrolimus
* Punctual plugs
* History of any of the following within previous six months:
* ocular trauma
* ocular infection, Ocular allergy
* History of any of the following within last 12 months:
* inflammatory corneal ulcer
* Herpetic eye infection
* or uveitis
* Ocular surgery

Systemic / non ophthalmic exclusion criteria:

•Known hypersensitivity to any of the components of the medical product under investigation or other study medication

Specific exclusion criteria for women:

* Pregnant or breast-feeding woman.
* Woman of childbearing potential (neither menopausal, nor hysterectomized, nor sterilized) not using effective contraception (i.e. hormonal contraceptives, intra-uterine device, contraceptive implant or condoms with spermicide)

Exclusion criteria related to general conditions

* Inability of patient to understand the investigation procedures and thus inability to give valid, informed consent.
* Non-compliant patient (e.g. not willing to attend the follow-up visits, way of life interfering with compliance)
* Participation in another clinical study or clinical investigation at the same time as the present investigation
* Participation to the present clinical investigation during the exclusion period of another clinical study
* Patient already included once in this clinical investigation
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited in University of Vienna
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Dryness score assessed by a VAS and Conjunctival hyperemia grading with Photographs (Efron) scale at week 12 | at week 12 versus baseline
  Scores will be determined using a 100 mm VAS on which 0 means "no feeling of eye dryness" and 100 means "most imaginable feeling of eye dryness".

IPD SHARING:
Plan to Share IPD: Undecided